CLINICAL TRIAL: NCT01150825
Title: Feasibility of High Frequency QRS Analysis in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BSP Biological Signal Processing Ltd. (Industry)
Responsible Party: Professor Doron Zahger, Soroka University Medical Center
Other Study IDs: ER_02_5023
Record Dates: First submitted 2010-06-10; First posted 2010-06-25 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Myocardial Infarction
Keywords: STEMI; NSTEMI; acute ischemia; non-invasive diagnosis; elevated troponin
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STEMI: Patients with ST segment elevation myocardial infarction, verified by elevated troponin levels
- NSTEMI: Patients with non-ST segment elevation myocardial infarction, verified by elevated levels of troponin

SUMMARY:
The primary objective of this study is to characterize the morphological patterns of high frequency QRS components (HFQRS) in patients with acute myocardial infarction (AMI), including STEMI and NSTEMI, compared to patients without AMI.

DETAILED DESCRIPTION:
Chest pain is one of the leading reasons of hospital emergency department (ED) visits worldwide. In the US, approximately 6 million people annually undergo evaluation in the ED for acute chest pain. Despite the wealth of knowledge available about acute coronary syndrome (ACS), this condition continues to be among the most difficult to predict or diagnose. Misdiagnoses may lead to discharge of patients with ACS, who should have been admitted as well as costly unnecessary hospitalizations of patients who do not have ACS.

More than 2/3 of the patients with ACS have unstable angina (UA) or non-ST-elevation myocardial infarction (NSTEMI). Conventional ECG has low sensitivity of less than 50% in diagnosing these conditions. As the initial ECG in the ED is often non-diagnostic in ACS patients, the diagnosis of ST-elevation myocardial infarction (STEMI) during its early stages may also be difficult.

Analysis of high-frequency QRS components (HFQRS), which quantifies changes in the depolarization phase of the cardiac cycle, has been previously reported to be a sensitive method for detection of demand ischemia. Preliminary studies have shown that HFQRS-derived indices can also identify supply ischemia caused by prolonged balloon occlusion, and transient ischemic episodes in patients with chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years (men and women)
* Time from onset of chest pain ≤ 12h
* AMI confirmed by biomarkers
* Clinical or electrocardiographic evidence of ischemia during recording
* Signed an informed consent

Exclusion Criteria:

* Prior MI
* Prior CABG
* pre-excitation syndrome (e.g. WP)
* Atrial Fibrillation or significant ventricular arrhythmia
* BBB, intraventricular conduction delay or QRS duration > 120 ms
* Implanted pacemaker or defibrillator
* Left-ventricular hypertrophy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with confirmed AMI in the intensive cardiac care unit (ICCU) of Soroka Medical Center (Beer Sheva, Israel), who are expected to undergo percutaneous coronary intervention (PCI) will be asked to participate in the study. These include both ST-elevation MI (STEMI) and non ST-elevation MI (NSTEMI) patients, with positive biomarkers and clear ongoing electrocardiographic or clinical evidence of ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Acute Myocardial Infarction | Prior to hospitalization release
  The primary end-point of the study is diagnosis of acute myocardial infarction, based on cardiac biomarkers, ECG changes clinical symptoms and coronary angiography.

SECONDARY OUTCOMES:
HFQRS analysis for detecting NSTEMI | Post data processing
  To evaluate the usefulness of HFQRS analysis in early detection of non-ST segment elevation myocardial infarction (NSTEMI).

CONTACTS AND LOCATIONS:
Overall Officials: Doron Zahger, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Derived] Amit G, Galante O, Davrath LR, Luria O, Abboud S, Zahger D. High-frequency QRS analysis in patients with acute myocardial infarction: a preliminary study. Ann Noninvasive Electrocardiol. 2013 Mar;18(2):149-56. doi: 10.1111/anec.12023. Epub 2012 Nov 22. PMID 23530485
- See also: Sponsor Website — http://www.bspmedical.com